CLINICAL TRIAL: NCT06814717
Title: A Phase 2a, Open-Label Study of the Safety, Tolerability, and Pharmacokinetics of a Single Dose of cP12 in Otherwise Healthy Adults With Up To and Including 5% Total Body Surface Area Thermal Burns
Brief Title: A Safety, Tolerability and Pharmacokinetic Study of cP12 in Adults With Up To 5% Total Body Surface Area Burns
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Neomatrix Therapeutics, Inc. (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NMT-cP12-201
Record Dates: First submitted 2025-01-17; First posted 2025-02-07 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-01

CONDITIONS: Thermal Burns

STUDY DESIGN:
Intervention Model Description: Safety study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label (Experimental): Six adult male or female subjects will receive a single administration of 0.01mg/kg of cP12.
  Interventions: Drug: cP12

INTERVENTIONS:
Drug: cP12 — cP12 is a novel fibronectin derived, 14-mer peptide

SUMMARY:
This is a Phase 2a, open-label, single-dose study to evaluate the safety, tolerability, and PK profile of cP12 in 6 male and female subjects with thermal burns of up to and including 5% TBSA. Enrolled subjects must have at least 1% TBSA deep partial-thickness burns.

Eligible subjects will receive a single administration of 0.01 mg/kg cP12. Vital signs, ECGs, and blood samples and urine samples will be obtained at screening and at several time points during the study for safety evaluation. Burn and pain assessments will be completed at specified times.

Subjects will remain at the clinical site for at least 6 hours post infusion for the purpose of safety monitoring and evaluation of other study assessments. Subsequent evaluations will be performed at the clinical site 3 (±1) days and 7 (±2) days after dosing.

Subjects will return to the clinical site 14 (±2) days after dosing for an End-of-Study visit.

DETAILED DESCRIPTION:
This is a Phase 2a, open-label, single-dose study to evaluate the safety, tolerability, and PK profile of cP12 in 6 male and female subjects with thermal burns of up to and including 5% TBSA. Enrolled subjects must have at least 1% TBSA deep partial-thickness burns. With the exception of the burns, subjects should be healthy and will be assessed to rule out smoke inhalation and other injuries. Vital signs prior to dosing must be stable and an electrocardiogram (ECG) must not show clinically significant abnormalities.

The target burn used in this study will be selected based on a burn classification description conducted prior to dosing with cP12. The selected burn must be deep partial-thickness and must not be a circumferential burn.

In the absence of burn-specific, validated assessment tools, NeoMatrix has developed scales to characterize the burn and surrounding tissues for this trial. Burn assessments will include erythema, capillary refill, blisters, and edema/swelling. In this trial, the target burn and all other burns of each subject will be assessed.

Eligible subjects will receive a single administration of 0.01 mg/kg cP12. Study drug will be administered over approximately 30 minutes by intravenous (IV) infusion with the subject in a supine position, and the infusion is to be initiated and completed within 2 to 12 hours after the burn has occurred. The subject is to remain in the supine position for 60 minutes from the start of study drug infusion (ie, during the 30-minute infusion and for 30 minutes after study drug infusion).

Vital signs, ECGs, and blood samples and urine samples will be obtained at screening and at several time points during the study for safety evaluation. Burn and pain assessments will be completed at specified times.

Subjects will remain at the clinical site for at least 6 hours post infusion for the purpose of safety monitoring and evaluation of other study assessments. Subsequent evaluations will be performed at the clinical site 3 (±1) days and 7 (±2) days after dosing.

Subjects will return to the clinical site 14 (±2) days after dosing for an End-of-Study visit.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 kg/m2 (inclusive) and body weight >/=50kg
* TBSA thermal burns up to and including 5%, with at least 1% deep partial- thickness burn
* Able to be infused with cP12 within 2 to 12 hours post burn
* Able to follow birth control requirements

Exclusion Criteria:

* Burns to the head, face and genitalia
* Smoke inhalation
* Active burn infection needing systemic antimicrobial treatment
* Full-thickness burn in the target burn
* Circumferential target burn
* Clinically significant laboratory abnormality or other clinical findings indicative of an exclusionary disease or medical history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events from dosing through follow-up | Day 1, Day 3 and Day 14
  Clinical safety labs will be collected
Incidence and severity of adverse events from dosing through follow-up | Day 1 (Baseline and 1hour, 6 hours postdose), Day 3 and Day 14
  Electrocardiograms will be performed
Incidence and severity of adverse events from dosing through follow-up | Baseline, Day 1 (2,5,15,30,60,90,120,240,360 minutes postdose), Day 3, Day 7 and Day 14
  Vital signs will be collected

SECONDARY OUTCOMES:
Investigate pharmacokinetic profile | Predose, 2,5,15,30,60,120 and 240 minutes post dose
  Blood samples will be analyzed for maximum plasma concentration (Cmax)
Investigate pharmacokinetic profile | Predose, 2,5,15,30,60,120 and 240 minutes post dose
  Blood samples will be analyzed for area under the plasma concentration (AUC) versus time curve
Investigate pharmacokinetic profile | Predose, 2,5,15,30,60,120 and 240 minutes post dose
  Blood samples will be analyzed for half-life (t1/2)
Investigate pharmacokinetic profile | Predose, 2,5,15,30,60,120 and 240 minutes post dose
  Blood samples will be analyzed for time to reach maximum plasma concentration (Tmax)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Shupp, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Medstar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No